CLINICAL TRIAL: NCT02899845
Title: Study of Improving Gait Parameters When Using a Cane in "Light Touch" Condition in Elderly People With and Without Walking Difficulties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-37; 2014-A01381-46 (Other: ANSM)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Disorders of Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- elderly people with walking difficulties (Experimental): subjects with proven gait disturbance and balance will be recruited from a walking speed test and a standardized geriatric assessment by a geriatrician
  Interventions: Other: postural task; Other: walk task
- elderly people without walking difficulties (Active Comparator): subjects with no gait disturbance and balance disorders will be recruited from a walking speed test and a standardized geriatric assessment, once the subjects with gait disturbance and balance disorders have been recruited in order to make a match on the age criterion
  Interventions: Other: postural task; Other: walk task

INTERVENTIONS:
Other: postural task
Other: walk task

SUMMARY:
This project aims to study the effect of haptic sensory information delivered at the hand using a cane in "light touch" or "light support" condition on postural stability and spatial and temporal gait parameters of elderly subjects with and without walking difficulties

ELIGIBILITY:
Inclusion Criteria:

* presence of gait disturbance or balance disorders defined by a geriatric assessment and / or a walking speed test

Exclusion Criteria:

* presence of acute problems or central or peripheral neurological severe sequelae
* occurrence of a recent fracture of the lower limbs or spinal fracture
* cognitive disorders
* presence of comorbidities: blindness, heart or severe respiratory failure, disabling osteoarthritis of the hands or legs, severe malnutrition, muscle atrophy, untreated orthostatic hypotension
* patients using a cane to a mechanical support

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
number of use of the cane | 12 mois

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No